CLINICAL TRIAL: NCT05408052
Title: Comparison of the Efficiency of Standard Epidural and Dural Puncture Epidural Analgesia Techniques Guided by Nociception Level Index in Open Gynecological Surgery Under General Anesthesia: a Prospective Randomized Double-Blind Study
Brief Title: Comparison of Standard Epidural and Dural Puncture Epidural Analgesia in Open Gynecological Surgery Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, Clinical Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/292
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Epidural (Active Comparator): Standard epidural technic will be applied before the anesthesia induction for perioperative analgesia
  Interventions: Procedure: Standart Epidural
- Dural Puncture Epidural (DPE) (Active Comparator): Dural Puncture Epidural technic will be applied before the anesthesia induction for perioperative analgesia
  Interventions: Procedure: Dural Puncture Epidural (DPE)

INTERVENTIONS:
Procedure: Dural Puncture Epidural (DPE) — Using the 18G Tuohy needle in the sitting position, the epidural space will be determined from the L3-L4 or L4-L5 space using the loss-of-resistance method After Dural puncture will be performed using a 25G Whitacre needle from the Tuohy needle to patients in the DPE group and free CSF flow will be observed, but no medication will be applied to the subarachnoid space. Afterwards, epidural catheter will be placed and when the catheter is fixed, a test dose of 3 mL will be administered through the catheter to check for intravascular or subarachnoid catheter placement.
  An epidural local anesthetic will be administered throughout the catheter for intraoperative analgesia at 0,1% (bupivacaine+fentanyl+ saline) concentration with the NoL monitor guidance.
  Arms: Dural Puncture Epidural (DPE)
Procedure: Standart Epidural — The neuraxial procedure will be performed in the sitting position using the 18G Tuohy needle, in the L3-L4 or L4-L5 range using the loss-of-resistance method.
  The epidural catheter will be placed so that it remains 4 to 5 cm in the epidural space. After the catheter is fixed, a test dose of 3 mL will be administered through the catheter to check for intravascular or subarachnoid catheter placement.
  An epidural local anesthetic will be administered throughout the catheter for intraoperative analgesia at 0,1% (bupivacaine+fentanyl+ saline) concentration with the NoL monitor guidance.
  Arms: Standard Epidural

SUMMARY:
The aim of this study is to compare the effectiveness of standard epidural and dural puncture epidural analgesia techniques used under NOL guidance.

The primary aim of this study was to evaluate the effect of NOL-guided antinociception on intraoperative total local anesthetic consumption during anesthesia.

The secondary aim is to compare onset time, analgesia duration time, hemodynamic parameters, time to first postoperative analgesic requirement, and postoperative side effects.

DETAILED DESCRIPTION:
This prospective randomized double-blind study was planned in 36 adult female patients aged 18-75 years, with ASA I-III, who underwent elective open gynecological surgery under general anesthesia with lower midline or Pfannenstiel incision after Ataturk University Medical Faculty Hospital ethics committee approval and written consent of the patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III physical condition
* patients aged between 18-75 years
* elective surgeries under general anesthesia for gynecological procedures
* lower midline or Pfannenstiel incision

Exclusion Criteria:

* patients with classical contraindications to neuraxial procedures,
* morbidly obese (body mass index > 40 kg / m2),
* pregnant and lactating women
* hypersensitive or allergic to local anesthetic agents,
* abuse of drugs or alcohol in the past 6 months.
* chronic opioid use before surgery,
* using chronic psychoactive drugs in the 90 days before surgery,
* patients with peripheral and central nervous system disease,
* preoperative hemodynamic compromise (patients with irregular sinus heart rhythm and pacemaker)
* patients using antimuscarinic, α2-adrenergic agonists, β1-adrenergic antagonists, antiarrhythmic agents,
* patients with diabetes, severe lung and significant liver disease with increased bilirubin,
* operations that will take less than 2 hours
* MAP >160 mmHg or <60 mmHg, heart rate >90 beats/min or <45 beats/min on the day of surgery
* patients who do not want to participate in the study will be excluded from the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to compare the total amount of epidural local anesthetics consumed during the intraoperative period | intraoperative period
  The primary outcome is to compare the total amount of epidural local anesthetics (mg) consumed during the intraoperative period

SECONDARY OUTCOMES:
Our secondary aim is to compare onset time | intraoperative period
  Our secondary aim is to compare onset time

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Dostbil, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)